CLINICAL TRIAL: NCT00520884
Title: A Pilot Study of Ghrelin in Healthy and Frail Older Women
Brief Title: Ghrelin in Healthy and Frail Older Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Anne Cappola, Associate Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IRB805400
Record Dates: First submitted 2007-08-23; First posted 2007-08-27 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-05

CONDITIONS: Frailty
Keywords: frailty; ghrelin; appetite; weight loss
MeSH Terms: conditions — Frailty; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy 70+ Women Placebo Infusion (Placebo Comparator): Healthy and Frail Women 70 and Older Receive a 3 hour Placebo Infusion of Saline administered in a stepwise fashion in amounts equivalent to the ghrelin infusion.
  Interventions: Other: Placebo Infusion -Healthy
- Frail 70+ Women Placebo Infusion (Placebo Comparator): Frail Women 70 and Older Receive a 3 hour Placebo Infusion of Saline administered in a stepwise fashion in amounts equivalent to the ghrelin infusion.
  Interventions: Other: Placebo Infusion - Frail
- Healthy 70+ Women Ghrelin Infusion (Active Comparator): Healthy Women 70 and Older are administered a 3 hour graded Ghrelin Infusion (the first hour of the ghrelin infusion a dose of 2.5 pmol/kg/min, increased to a dose of 5.0 pmol/kg/min for one hour, and then increased to the dose of 10 pmol/kg/min for the final hour of the infusion).
  Interventions: Drug: Ghrelin Infusion - Healthy
- Frail 70+ Women Ghrelin Infusion (Active Comparator): Frail Women 70 and Older are administered a 3 hour graded Ghrelin Infusion (the first hour of the ghrelin infusion at a dose of 2.5 pmol/kg/min, increased to a dose of 5.0 pmol/kg/min for one hour, and then increased to the dose of 10 pmol/kg/min for the final hour of the infusion).
  Interventions: Drug: Ghrelin Infusion - Frail

INTERVENTIONS:
Drug: Ghrelin Infusion - Healthy — At time 0, a graded infusion of Ghrelin of 2.5, 5.0, and 10.0 pmol/kg/min infused in one of the IV sites for 60 minutes each, totalling 180 minutes when the infusion will be stopped.
  Other Names: Healthy Older Women Receiving
  Arms: Healthy 70+ Women Ghrelin Infusion
Drug: Ghrelin Infusion - Frail — At time 0, a graded infusion of Ghrelin of 2.5, 5.0, and 10.0 pmol/kg/min will be infused in one of the IV sites for 60 minutes each, totalling 180 minutes when the infusion will be stopped.
  Other Names: Frail Older Women Receiving
  Arms: Frail 70+ Women Ghrelin Infusion
Other: Placebo Infusion -Healthy — At time 0, an infusion of saline will be started in one of the IV sites (an equivalent amount to compare to the Ghrelin infusion) and will be infused in a stepwise fashion continued until 180 minutes, when the infusion will be stopped.
  Other Names: Healthy Older Women Receiving
  Arms: Healthy 70+ Women Placebo Infusion
Other: Placebo Infusion - Frail — At time 0, an infusion of saline will be started in one of the IV sites (an equivalent amount to compare to the Ghrelin infusion) and will be infused in a stepwise fashion continued until 180 minutes, when the infusion will be stopped.
  Other Names: Frail Older Women Receiving
  Arms: Frail 70+ Women Placebo Infusion

SUMMARY:
The purpose of this research study is to see if giving women a hormone called "ghrelin" will increase levels of growth hormone in the blood and increase appetite. Ghrelin is a naturally occurring hormone that is produced mostly by the stomach and causes secretion of another hormone called growth hormone. It also increases short-term appetite and may lower the amount of inflammation in the body.

Some people lose their appetite as they age and have unintentional weight loss. This may be caused by a break in the communication between the stomach and the brain. We are particularly interested in seeing if there is a difference in the effects of ghrelin in older women who have lost weight recently without wanting to and those who have not.

DETAILED DESCRIPTION:
Five community-dwelling women aged 70 or over with unintentional weight loss of >5% in the prior year plus at least 2 of the 4 remaining Fried criteria for frailty and five healthy women without any frailty criteria were enrolled. Women with conditions that can cause weight loss or taking an appetite stimulant or corticosteroids were excluded. Each woman completed two 180 minute infusions, one week apart, assigned randomly: a graded ghrelin infusion of 2.5, 5.0, and 10.0 pmol/kg/min for 60 minutes each and an equivalent placebo (saline) infusion. A meal of standardized composition was provided after each infusion and intake quantified. Samples were collected every 30 minutes for growth hormone (GH), and total and active ghrelin. Additional samples were collected every 60 minutes for glucose, insulin, free fatty acids, leptin, adiponectin, resistin, glucagon-like peptide-1 receptor agonists (GLP-1), and cortisol. Adverse events were collected during the infusion and by telephone 24 hours later. Non-parametric methods were used to compare differences in response to the ghrelin and placebo infusions 1) in all women and 2) between frail and healthy women.

ELIGIBILITY:
Inclusion Criteria:

Frail group:

* Women aged 70 or greater
* Able to give informed consent
* Undiagnosed weight loss (>5% over the previous year)
* Two of the following four criteria (from Fried L et al, 2001): low grip strength, slow walking speed, subjective exhaustion, low levels of physical activity

Healthy group:

* Women aged 70 or greater
* Able to give informed consent
* None of the frailty criteria

Exclusion Criteria:

* Prior diagnosis of Parkinson's Disease
* History of cerebrovascular accident with residual hemiparesis
* Hospitalization for treatment of vascular disease (including, coronary heart disease, cerebrovascular disease, peripheral vascular disease) in the past 6 months
* Congestive heart failure
* Rheumatoid arthritis or other inflammatory conditions
* Depression (defined as a score of >11 on the Geriatric Depression Questionnaire)
* History of cancer requiring treatment in the past 5 years, with the exception of cancers which have been cured, or, in the opinion of the investigator, carry a good prognosis
* Cognitive deficit as defined by a Folstein Mini Mental State Exam score < 18/30
* Current use of corticosteroids or immune-modulating agents other than topical, ophthalmic, and inhaled preparations, in past 3 months
* Diabetes mellitus
* Thyroid stimulating hormone (TSH) measured as <0.5 U/L or greater than 10 U/L. If participant is taking replacement thyroid hormone, they should be on a stable dose for at least 2 months
* History of liver disease or abnormal liver function tests (LFTs > 2x upper limit of normal)
* Renal insufficiency (serum creatinine ≥ 1.4 mg/dL).
* Hemoglobin < 11g/dL
* History of surgery within the last 30 days.
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study
* Participation in an investigational drug study within 6 weeks prior to screening visit
* Self reported history of HIV disease
* Hospitalization for chronic obstructive pulmonary disease or asthma in the past 3 months
* History of alcohol abuse as defined as any one of the following:

  1) average consumption of 3 or more alcohol containing beverages daily; 2) consumption of 7 or more alcoholic beverages within a 24 hr period in the past 12 months; or 3) clinical assessment of alcohol dependence based on two or more positive responses to an alcoholism questionnaire (if confirmed by further probing) or on other evidence available to clinic staff. If any of these exclusion criteria are met, the subject may still be considered eligible if, after an explanation of the importance of limiting alcohol intake during the study, the clinic staff believes that the volunteer can and will limit future alcohol intake to acceptable levels.
* History of gastrectomy
* Current therapy with an appetite stimulant, i.e. medroxyprogesterone acetate, within the last 6 weeks.
* Weight >85 kg

Min Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne R Cappola, MD, ScM, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Clinical and Translational Research Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventeen women were screened. Ten qualified - five had unintentional weight loss of >5% in the prior year plus at least 2 out of the 4 remaining Fried criteria for frailty and five healthy women without any frailty criteria. Women with conditions that can cause weight loss or taking an appetite stimulant or corticosteroids were excluded.
Groups:
- Healthy Participants, Ghrelin First, Then Saline: Healthy participants, ghrelin first, then saline
- Healthy Participants, Saline First, Then Ghrelin: Healthy participants, saline first, then ghrelin
- Frail Participants, Ghrelin First, Then Saline: Frail participants, ghrelin first, then saline
- Frail Participants, Saline First, Then Ghrelin: Frail participants, saline first, then ghrelin
Period: Overall Study
Arm/Group | Healthy Participants, Ghrelin First, Then Saline | Healthy Participants, Saline First, Then Ghrelin | Frail Participants, Ghrelin First, Then Saline | Frail Participants, Saline First, Then Ghrelin
Started | 3 | 2 | 2 | 3
Completed (Crossover study, randomized in two strata) | 3 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy; Frail: Receiving Placebo at one visit/Ghrelin at other visit
- Total: Total of all reporting groups
Arm/Group | Healthy | Frail | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Full Range); unit: years] | 80.6 [73 to 94] | 80.0 [75 to 85] | 80.3 [73 to 94]
Sex/Gender, Customized [Number; unit: participants] | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Kilocalories Consumed
Description: Kilocalorie consumption from meal of standardized composition during the visit when infusion complete
Time Frame: After infusion
Population: Per protocol, primary analysis combined healthy and frail groups. The study was not powered to make statistical comparisons between the healthy and frail groups. Therefore, we are providing combined data per our protocol.
Measure: Mean (Standard Deviation); unit: Kilocalorie
Groups:
- Saline Infusion; Ghrelin Infusion: Saline infusion in combined healthy and frail groups
Arm/Group | Saline Infusion | Ghrelin Infusion
Number analyzed (Participants) | 10 | 10
Kilocalorie | 412 (151) | 553 (151)

2. Primary Outcome: Max Change Growth Hormone
Description: Maximum growth hormone level change from baseline to 180 minutes
Time Frame: 180 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ghrelin Infusion: Ghrelin infusion in combined healthy and frail groups
Arm/Group | Saline Infusion | Ghrelin Infusion
Number analyzed (Participants) | 10 | 10
ng/mL | 0.33 (1.44) | 14.24 (8.49)

3. Primary Outcome: Max Change Total Ghrelin
Description: Maximum total ghrelin change from baseline to 180 minutes
Time Frame: 180 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Saline Infusion | Ghrelin Infusion
Number analyzed (Participants) | 10 | 10
pg/mL | -68.6 (90.6) | 1803.2 (714.8)

4. Primary Outcome: Max Change Active Ghrelin
Description: Active ghrelin change from baseline to 180 minutes. Active ghrelin=acylated ghrelin.
Time Frame: 180 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Saline Infusion | Ghrelin Infusion
Number analyzed (Participants) | 10 | 10
pg/mL | -9.1 (20.4) | 845.4 (448.3)

ADVERSE EVENTS:
Time Frame: 1 week after each infusion
Groups:
- Placebo: Healthy and frail participants had a study visit in which they received placebo (saline) infusion
- Ghrelin: Healthy and frail participants had a study visit in which they received ghrelin infusion
Arm/Group | Placebo | Ghrelin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Ghrelin (N=10)
sensation of warmth (General disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes